CLINICAL TRIAL: NCT05713461
Title: Effects of a Physical Exercise Program Adapted to People With Obesity on Health Indicators and Quality of Life.
Brief Title: Physical Exercise in Obesity for Health and Quality of Life.
Acronym: OBEFYSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pablo de Olavide (Other)
Collaborators: University of Seville (Other)
Responsible Party: Principal Investigator, José Antonio González Jurado, PhD, Universidad Pablo de Olavide
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UPO-1381609
Record Dates: First submitted 2023-01-07; First posted 2023-02-06 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Overweight and Obesity; Overweight or Obesity
Keywords: lipoinflammation; metabolic syndrome; training; overweight; sedentary lifestyle
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: To compare the effects of an interval training program in obese women with metabolic syndrom vs obese women without metabolic syndrom
Who Masked: Participant, Investigator
Masking Description: Participants do not know if they have metabolic syndrom Physical training supervisors do not know if participants have metabolic syndrom
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obese women without metabolic syndrome (Experimental): Women with obesity and without metabolic syndrome
  Interventions: Behavioral: exercise training program; Behavioral: Feeding training
- obese women with metabolic syndrome (Experimental): Women with obesity and with metabolic syndrome
  Interventions: Behavioral: exercise training program; Behavioral: Feeding training

INTERVENTIONS:
Behavioral: exercise training program — Adapted Interval Training Intervention, three days a week, 10 weeks.
  Warm-up 10': Joint mobility and cardiovascular activation
  Main part:
  Resistance training circuit for strengthening the main muscle groups.
  Cool down Flexibility and CORE
  Other Names: interval training program
Behavioral: Feeding training — Two workshops on healthy eating habits (Week 1 and week 5). Food Frequency Questionnaires (weekly). Feedback weekly. Mediterranean Diet Adherence Screener (MEDAS). The dietary intervention will be based on the nutritional recommendations based on the Mediterranean diet, according to the evidence from the PREDIMED trial.

SUMMARY:
This project aims to develop an intervention on healthy habits based on physical exercise and nutritional education in people with obesity.

It is accepted that exercise and nutrition are keys to controlling body weight. People with obesity frequently present with metabolic syndrome and a low-grade inflammatory state.

It is not known what should be the most effective training load/dose (duration, intensity, type of exercise) to improve health indicators related to metabolic syndrome and lipo-inflammation, and body composition in people with obesity.

A large-scale randomized controlled trial (RCT) will be essential to better understand the type and characteristics of training load/dose most effective in counteracting the detrimental effects of obesity.

The aim of this trial in 50 obese women was to answer the following questions:

* Does the training program improve physical fitness?
* Does the training program improve body composition?
* Does the training program improve the state of chronic low-grade inflammation?
* Does the training program improve the quality of life and perceived health?
* Do people with obesity and metabolic syndrome respond in the same way to training?
* what is the effect of four weeks of detraining?

DETAILED DESCRIPTION:
A female single group, 2-armed ( people with obesity and metabolic syndrome vs people with obesity without metabolic syndrome), investigator-blinded, trial.

The study will last 17 weeks. Week 1 (testing 1: pretest); weeks 2-11 (Intervention: interval training program); week 12 (testing 3: postest); weeks 13-16 (detraining period); week 17 (testing 3: detraining test)

Participants will be allocated (1:1) regarding metabolic syndrome Behavioural: exercise training program Adapted Interval Training Intervention, three days a week, 10 weeks.

Warm-up ≃ 10': Joint mobility and cardiovascular activation.

Main part ≃ 45 min.:

Resistance training circuit for strengthening the main muscle groups.

* Shoulder muscles
* Pectoral muscles
* Knee Flexor-extensor muscles
* hip flexor extensor muscles Between 50-70% 1 RM (estimated). Repetitions 1-2 RIR (Repetition in Reserve). Load Intensity was controlled through RPE (OMNI-RES Scale) between 7-8 out of 10.

The training load will increase while maintaining the same intensity.

Cool down ≃ 5' Flexibility and CORE

Behavioural: Feeding training Two workshops on healthy eating habits (Week 1 and week 5). Food Frequency Questionnaires (weekly). Feedback weekly Mediterranean Diet Adherence Screener (MEDAS) The dietary intervention will be based on the nutritional recommendations based on the Mediterranean diet, according to the evidence from the PREDIMED trial.

ELIGIBILITY:
Inclusion Criteria:

* The recruitment of participants would be carried out through advertising in the press, social networks, and electronic media.

Main inclusion criteria

* Sex: Female
* Caucasian
* Age. women from 35 years to 65 years.
* BMI: >29
* Abdominal perimeter: >90 cm women
* No known Diabetes
* No known cancer
* No Known lung disease
* No known cardiovascular disease
* No known thyroid disease
* No known liver disease
* No known autoimmune disease
* No other endocrine disorder causes obesity
* No current treatment with anti-obesity medication
* No current treatment with anti-inflammatory medication
* No weight loss of > 5kg within the last 6 months
* No diagnosis of depression or treatment with anti-depressive medication, ongoing or within the last three months before enrolment
* No diagnosis of psychiatric disorder or treatment with antipsychotic medication
* No history of suicidal behavior or ideations within the last three months before enrolment
* No previous surgical treatment for obesity
* Not pregnant/considering pregnancy
* No functional impairments that prevent the performance of intensive exercise
* Declare a sedentary lifestyle ((< 1,5 hours of structured physical activity per week at moderate intensity)
* No participation in other research intervention studies
* Signed informed consent.

Exclusion Criteria:

* Diagnosis of pathology that involves an inflammatory process in the last year.
* Objective findings that contraindicate participation in intensive exercise
* The language barrier, mental incapacity, unwillingness or inability to understand the instruction of the study
* Not completing 75% of the training sessions

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in low-grade chronic inflammation | from baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  Plasma levels of inflammatory and lipoinflammatory markers
  Multiplex Quantitative measurement of 40 human adipokines in plasma (cytokine antibody arrays (pg/ml) :
  1. Adiponectin
  2. Adipsin
  3. AgRP
  4. ANGPTL4
  5. BDNF
  6. Chemerin
  7. CRP
  8. GH
  9. IFNg
  10. IGFBP-1
  11. IGFBP-2
  12. IGF-I
  13. IL-10
  14. IL-12p40
  15. IL-12p70
  16. IL-1b
  17. IL-1ra
  18. IL-6
  19. IL-8
  20. Insulin
  21. Leptin
  22. Lipocalin-2
  23. MSPa
  24. OPG
  25. PAI-1
  26. PDGF-BB
  27. Pepsinogen 1
  28. Pepsinogen 2
  29. Procalcitonin
  30. Prolactin
  31. RANTES
  32. RBP4
  33. Resistin
  34. SAA
  35. TGFb1
  36. TSP-1
  37. TNF RI
  38. TNF RII
  39. TNFa
  40. VEGF
Change in body composition | from baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  Body composition by DEXA. Main body composition components:
  * Body Fat Mass (g)
  * Body Lean Mass (g)
  * Body Bone mineral content (g)
  * Body Total mass (g)
  * Estimated Visceral Adipose Tissue (g)
  * BMI: kg/m^2
Change in physical fitness (resistance; muscular strength) | from baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  * Maximum dynamic strength of the upper body (bench press; kg)
  * Lower body maximal dynamic strength (leg press; kg)
  * Grip maximal isometric strength (handgrip: kg)
Change in physical fitness (aerobic power; VO2max) | From baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  Aerobic power. VO2 max. (estimated from the 6-minute walk test; ml/kg/min)
Change in physical fitness (Coordination; balance) | From baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  Balance test one leg (seconds)
Change in perceived health and perceived quality of life | from baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  perceived health by questionnaire (SF-12). The SF-12 response options are Likert-type scales that assess intensity or frequency.
  The number of response options ranges from three to six, depending on the item, and each question receives a value that is later transformed into a scale from 0 to 100.
Change in healthy eating habits | from baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  Mediterranean Diet Adherence Screener (MEDAS). MEDAS consists of 12 questions on food consumption frequency and 2 questions on food intake habits considered characteristic of the Spanish Mediterranean diet. Each question was scored 0 or 1.

SECONDARY OUTCOMES:
Change eating habits | Every week, from baseline (0 weeks) to follow-up (10 weeks)
  Food Frequency Questionnaires (weekly). Recording the frequency of food consumption per week
Change in Biochemistry Determinations In Plasma (lipidic profile) | From baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  LIPIDIC PROFILE Total Cholesterol (mg/dl) HDL Cholesterol (mg/dl) LDL Cholesterol (mg/dl) Triglycerides (mg/dl)
Change in Biochemistry Determinations In Plasma (glucose metabolism) | From baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  Glycosylated Hemoglobin A1c (%) Insulin (uU/ml) Glucose (mg/dl) Insulin Resistance. HOMA-IR = (fasting insulin (uU/ml) * fasting glucose (mg/dl)) / 405
Change in Biochemistry Determinations In Plasma (Enzymes of fatigue or muscular damage) | From baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  ENZYMES (Fatigue or muscular damage) Creatine Kinase (UI/L) Transaminases (GOT/AST, GPT/ALT, GGT; UI/L ) C-Reactive Protein (mg/l)
Change in Biochemistry Determinations In Plasma (protein metabolism) | From baseline ( 0 weeks) to follow-up (10 weeks) and detraining effects (after 4 weeks sedentary lifestyle)
  PROTEIN METABOLISM Uric Acid (mg/dl) Urea (mg/dl) Creatinine (mg/dl) Bilirubin (mg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Gonzalez-Jurado, PhD, Principal Investigator — Universidad Pablo de Olavide de Sevilla
Locations (1):
- CIRFD Universidad Pablo de Olavide, Seville, Spain